CLINICAL TRIAL: NCT03886935
Title: Metabolic Remodeling in Fontan Patients: a Metabolomics Study
Brief Title: Metabolic Remodeling in Fontan Patients
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Biocrates Life Sciences AG, Innsbruck, Austria (Unknown); Tiroler Wissenschaftsförderung (Unknown)
Responsible Party: Sponsor
Other Study IDs: 201810011837
Record Dates: First submitted 2019-03-11; First posted 2019-03-22 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2017-01

CONDITIONS: Congenital Heart Disease; Metabolism Disorder
MeSH Terms: conditions — Heart Defects, Congenital; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fontan patients: The serum of Fontan patients is compared to the serum of healthy biventricular controls (Metabolomics)
  Interventions: Diagnostic Test: Metabolomics
- Healthy biventricular controls: The serum of Fontan patients is compared to the serum of healthy biventricular controls (Metabolomics)
  Interventions: Diagnostic Test: Metabolomics

INTERVENTIONS:
Diagnostic Test: Metabolomics

SUMMARY:
Assessment of metabolic alterations in adult Fontan patients with a dominant left ventricle with the help of serum examinations (Metabolomics). The aim is to find a tool for the completion of the (semi-)invasive monitoring of Fontan hemodynamics.

DETAILED DESCRIPTION:
Patients who are born with just one single heart chamber need to undergo surgical therapy allowing the single heart chamber to pump the blood into the systemic circulation and allowing the blood to flow passively to the lungs (Fontan circulation). Regular ultrasound, cardiopulmonary exercise testing, and invasive diagnostic tools (catheterization, general anaesthesia needed) are necessary to early find out cardiac, vascular, or circulatory impairment. It is still very difficult to diagnose and therapy failure of this Fontan system early enough.

It is reported that in patients with a failing two-chambered heart, the energy source for the heart and the body in general switches from the use of lipids to the use of sugar and ketone bodies. First studies show decreased concentrations of membrane lipids in Fontan patients with a left dominant ventricle, and the energy metabolism has not been focused yet in those patients.

The investigators hypothesize that there are differences in the pattern of the structural metabolism in adult Fontan patients with a left-dominant vs. a right-dominant ventricle. Furthermore the investigators hypothesize that there are alterations in the energy metabolism in adult Fontan patients in comparison to healthy two-chambered controls, and that those alterations correlate with the grade of impairment of cardiopulmonary function.

With the help of a special biochemical examination (mass spectrometry-based Metabolomics study) blood of Fontan patients will be analyzed, and the results will be correlated with the results of ultrasound and cardiopulmonary exercise testing. The aim of this study is to establish sensitive blood markers indicating cardiac, vascular, circulatory or further organ dysfunction in Fontan patients. This should allow optimal Fontan system monitoring with an optimal timing of an additional invasive diagnostic catheterization and of nutritional, medical or interventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fontan circulation (right systemic ventricle), biventricular heart with heart failure resp.
* ≥ 18 years
* Written informed consent of patients
* 8 hours fasting period before blood sample

Exclusion Criteria:

Intake of medication directly affecting metabolic (e.g. metabolism of lipids (statine)) or hemodynamic state (e.g. beta-blockers, sildenafil) (other than angiotensin converting enzyme (ACE)-inhibitors and anticoagulation therapy)

* Cachectic disease
* Non-congestive hepatic or renal dysfunction
* (Inherited) metabolic disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥ 18 years with a Fontan circulation with a dominant left ventricle.
  Controls: age- and sex-matched healthy biventricular controls ≥ 18 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Metabolism of lipids | blood sampling at one single point of time (baseline/day 1) in the context of a planned patient presentation at the pediatric cardiology outpatient clinic (without assessment of changes)
  Measurement of the serum concentration of the extended metabolism of lipids using the technique of Metabolomics (AbsoluteIDQ p180 kit, Biocrates Life Sciences AG, Innsbruck, Austria)
Metabolism of amino acids and related compounds | blood sampling at one single point of time (baseline/day 1) in the context of a planned patient presentation at the pediatric cardiology outpatient clinic (without assessment of changes)
  Measurement of the serum concentration of the extended metabolism of lamino acids using the technique of Metabolomics (AbsoluteIDQ p180 kit, Biocrates Life Sciences AG, Innsbruck, Austria)
Metabolism of carbohydrates | blood sampling at one single point of time (baseline/day 1) in the context of a planned patient presentation at the pediatric cardiology outpatient clinic (without assessment of changes)
  Measurement of the serum concentration of the extended metabolism of carbohydrates using the technique of Metabolomics (AbsoluteIDQ p180 kit, Biocrates Life Sciences AG, Innsbruck, Austria)
Metabolism of ketone bodies | blood sampling at one single point of time (baseline/day 1) in the context of a planned patient presentation at the pediatric cardiology outpatient clinic (without assessment of changes)
  Measurement of the serum concentration of ketone bodies using the technique of Metabolomics (AbsoluteIDQ p180 kit, Biocrates Life Sciences AG, Innsbruck, Austria)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Karall, Prof., Principal Investigator — Medical University of Innsbruck

IPD SHARING:
Plan to Share IPD: No
Participant data will be available only to the head of the study (Dr. Miriam Michel) (Excel- and SPSS-files)

REFERENCES:
- [Derived] Michel M, Salvador C, Wiedemair V, Adam MG, Laser KT, Dubowy KO, Entenmann A, Karall D, Geiger R, Zlamy M, Scholl-Burgi S. Method comparison of HPLC-ninhydrin-photometry and UHPLC-PITC-tandem mass spectrometry for serum amino acid analyses in patients with complex congenital heart disease and controls. Metabolomics. 2020 Dec 15;16(12):128. doi: 10.1007/s11306-020-01741-8. PMID 33319318
- [Derived] Michel M, Dubowy KO, Zlamy M, Karall D, Adam MG, Entenmann A, Keller MA, Koch J, Odri Komazec I, Geiger R, Salvador C, Niederwanger C, Muller U, Scholl-Burgi S, Laser KT. Targeted metabolomic analysis of serum phospholipid and acylcarnitine in the adult Fontan patient with a dominant left ventricle. Ther Adv Chronic Dis. 2020 Apr 27;11:2040622320916031. doi: 10.1177/2040622320916031. eCollection 2020. PMID 32426103